CLINICAL TRIAL: NCT03909165
Title: A Phase 4 Double-blinded, Randomized, Active Comparator-controlled Clinical Trial to Study the Efficacy, Safety, and Pharmacokinetics of Sugammadex (MK-8616) for Reversal of Neuromuscular Blockade in Pediatric Participants Aged Birth to <2 Years
Brief Title: Efficacy, Safety, and Pharmacokinetics of Sugammadex (MK-8616) for Reversal of Neuromuscular Blockade in Pediatric Participants Aged Birth to <2 Years (MK-8616-169)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8616-169; MK-8616-169 (Other: MSD Protocol Number); 2017-000693-11 (EudraCT Number)
Record Dates: First submitted 2019-04-08; First posted 2019-04-09 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate; Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A will be open-label, while Part B will be double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A. Sugammadex 2 mg/kg (Experimental): Participants received a single intravenous (IV) bolus of sugammadex at 2 mg/kg for moderate NMB reversal.
  Interventions: Drug: Sugammadex 2 mg/kg
- Part A. Sugammadex 4 mg/kg (Experimental): Participants received a single IV bolus of sugammadex at 4 mg/kg for deep NMB reversal.
  Interventions: Drug: Sugammadex 4 mg/kg
- Part B. Sugammadex 2 mg/kg (Experimental): Participants received a single IV bolus of sugammadex at 2 mg/kg for moderate NMB reversal.
  Interventions: Drug: Sugammadex 2 mg/kg
- Part B. Sugammadex 4 mg/kg (Experimental): Participants received a single IV bolus of sugammadex at 4 mg/kg for deep NMB reversal.
  Interventions: Drug: Sugammadex 4 mg/kg
- Part B. Neostigmine (Active Comparator): Participants received a single IV bolus containing neostigmine (50 μg/kg; up to 5 mg maximum dose) in combination with either glycopyrrolate (10 μg/kg) or atropine sulfate (20 μg/kg) based on availability and/or contraindications, for moderate NMB reversal.
  Interventions: Drug: Neostigmine + Glycopyrrolate; Drug: Neostigmine + Atropine

INTERVENTIONS:
Drug: Sugammadex 2 mg/kg — For moderate NMB reversal, a single IV bolus of sugammadex (2 mg/kg) will be given after final dose of neuromuscular blocking agent (NMBA; rocuronium or vecuronium) and within 2 minutes of the reappearance of a second twitch (T2) in response to train-of-four (TOF) stimulations.
  Other Names: MK-8616
  Arms: Part A. Sugammadex 2 mg/kg; Part B. Sugammadex 2 mg/kg
Drug: Sugammadex 4 mg/kg — For deep NMB reversal, a single IV bolus of sugammadex (4 mg/kg) will be given after final dose of NMBA (rocuronium or vecuronium) and within 2 minutes of detection of a target of 1 to 2 post-tetanic counts and no response to TOF stimulations (TOF=0).
  Other Names: MK-8616
  Arms: Part A. Sugammadex 4 mg/kg; Part B. Sugammadex 4 mg/kg
Drug: Neostigmine + Glycopyrrolate — For moderate NMB reversal, a single i.v. bolus containing both neostigmine (50 μg/kg; up to 5 mg maximum dose) as well as glycopyrrolate (10 μg/kg) will be given after final dose of NMBA (rocuronium or vecuronium) and within 2 minutes of the reappearance of T2 in response to TOF stimulations.
  Arms: Part B. Neostigmine
Drug: Neostigmine + Atropine — For moderate NMB reversal, a single i.v. bolus containing both neostigmine (50 μg/kg; up to 5 mg maximum dose) as well as atropine (20 μg/kg) will be given after final dose of NMBA (rocuronium or vecuronium) and within 2 minutes of the reappearance of T2 in response to TOF stimulations.
  Arms: Part B. Neostigmine

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics (PK) of sugammadex (MK-8616) for reversal of both moderate and deep neuromuscular blockade (NMB) in pediatric participants aged birth to <2 years. The primary hypothesis of this study is that sugammadex is superior to neostigmine in reversing moderate NMB as measured by time to neuromuscular recovery.

DETAILED DESCRIPTION:
This trial will be conducted in two parts: Part A and Part B. In Part A, PK sampling will be conducted to identify the pediatric dose providing sugammadex exposure comparable to the next oldest age cohort. For Part B participants, the efficacy of sugammadex (i.e. neuromuscular recovery / time to extubation) will be assessed. Further, safety analyses will be conducted in both Parts A and B. Following completion of Part A, an interim analysis (IA) of the PK and safety data will be performed. Once the appropriate doses are confirmed and safety data is assessed for the 2 doses of sugammadex, then Part B will commence.

ELIGIBILITY:
Inclusion Criteria:

* Categorized as American Society of Anesthesiologists (ASA) Physical Status Class 1, 2, or 3.
* Has a planned non-emergent surgical procedure or clinical situation (e.g., intubation) that requires moderate or deep NMB with either rocuronium or vecuronium.
* Has a surgical procedure or clinical situation that would allow neuromuscular monitoring techniques to be applied for neuromuscular transmission monitoring.
* Is male or female, between birth and <2 years of age.

Exclusion Criteria:

* Is a preterm infant or neonate <36 weeks gestational age at birth.
* Has any clinically significant condition or situation (e.g., anatomical malformation that complicates intubation) other than the condition requiring the use of NMBA that, in the opinion of the investigator, would interfere with the trial evaluations or optimal participation in the trial.
* Has a neuromuscular disorder that may affect NMB and/or trial assessments.
* Is dialysis-dependent or has (or is suspected of having) severe renal insufficiency.
* Has or is suspected of having a family or personal history of malignant hyperthermia.
* Has or is suspected of having an allergy to study treatments or its/their excipients, to opioids/opiates, muscle relaxants or their excipients, or other medication(s) used during general anesthesia.
* Is expected to require mechanical ventilation after the procedure.
* Has received or is planned to receive toremifene and/or fusidic acid via IV administration within 24 hours before or within 24 hours after administration of study treatment.
* Use of medication expected to interfere with study treatments given in this trial.
* Has been previously treated with sugammadex or has participated in a sugammadex clinical trial within 30 days of signing the informed consent form of this current trial.
* Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 30 days of signing the informed consent/assent for this current trial.

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (39):
- United States (7):
  - Lucille Packard Children's Hospital ( Site 3008), Palo Alto, California
  - Variety Children's Hospital D.B.A. Nicklaus Children's Hospital ( Site 3019), Miami, Florida
  - OU Medical Center ( Site 3005), Oklahoma City, Oklahoma
  - The Children's Hospital of Philadelphia ( Site 3021), Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh UPMC ( Site 3017), Pittsburgh, Pennsylvania
  - McGovern Medical School at UT Health/ Memorial Hermann ( Site 3014), Houston, Texas
  - University of Vermont Medical Center ( Site 3013), Burlington, Vermont
- Australia (3):
  - The Children s Hospital at Westmead ( Site 3805), Westmead, New South Wales
  - Queensland Children s Hospital ( Site 3806), South Brisbane, Queensland
  - Royal Childrens Hospital Melbourne ( Site 3801), Parkville, Victoria
- Belgium (3):
  - Universitaire Ziekenhuis Antwerpen - UZA ( Site 3200), Edegem, Antwerpen
  - UZ Brussel ( Site 3201), Brussels, Bruxelles-Capitale, Region de
  - UZ Leuven - Campus Gasthuisberg ( Site 3202), Leuven, Vlaams-Brabant
- Brazil (3):
  - Hospital Pequeno Principe ( Site 3826), Curitiba, Paraná
  - Hospital Tacchini ( Site 3827), Bento Gonçalves, Rio Grande do Sul
  - Instituto da Crianca do Hospital das Clinicas-FMUSP ( Site 3825), São Paulo
- Rigshospitalet ( Site 3250), Copenhagen, Capital Region, Denmark
- New Childrens Hospital ( Site 3750), Helsinki, Uusimaa, Finland
- C.H.R.U. de Lille. Hopital Jeanne de Flandres ( Site 3304), Lille, Nord, France
- Unidad de Cirugía Cardiovascular ( Site 4126), Guatemala City, Guatemala
- Hungary (2):
  - Szegedi Tudomanyegyetem ( Site 4201), Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont ( Site 4200), Debrecen
- Malaysia (3):
  - Sarawak General Hospital ( Site 3877), Kuching, Sarawak
  - Women and Children Hospital Kuala Lumpur (Hospital Tunku Azizah) ( Site 3875), Kuala Lumpur
  - University Malaya Medical Centre. ( Site 3876), Kuala Lumpur
- Mexico (2):
  - Hospital General de Zona No. 1 ( Site 4153), Ciudad de Villa de Álvarez, Colima
  - Centenario Hospital Miguel Hidalgo-Pediatrics Department ( Site 4152), Aguascalientes
- Netherlands (4):
  - Radboud University Medical Center ( Site 4226), Nijmegen, Gelderland
  - Erasmus University Medical Center ( Site 4225), Rotterdam, South Holland
  - University Medical Center Groningen ( Site 4227), Groningen
  - Wilhelmina Kinderziekenhuis ( Site 4228), Utrecht
- Instituto Nacional Cardiovascular Incor ( Site 3928), Lima, Peru
- Russia (7):
  - Scientific Research Institute Complex Problems Cardiovascular Disease ( Site 4288), Kemerovo, Kemerovo Oblast
  - NMRC Obstetrics Gynecology and Perinatology n.a. V.I. Kulakov ( Site 4287), Moscow, Moscow
  - Pediatric Hematology Oncology and Immunology Centre n.a. D.Rogachev. ( Site 4275), Moscow, Moscow
  - Children City Clinical Hospital 13 n.a N.F.Filatov ( Site 4285), Moscow, Moscow
  - Children City Clinical Hospital #9 n.a. G.N.Speransky ( Site 4290), Moscow, Moscow
  - Scientific-Research Clinical Pediatric Institution n.a. Veltischev ( Site 4276), Moscow, Moscow
  - St.Petersburg State Pediatric Medical University ( Site 4281), Saint Petersburg, Sankt-Peterburg

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Mensah-Osman E, Mukai Y, Wang A, Matuszczak M, Saldien V, Leibensperger H, Speek M, Locco A, Wrishko R, Gee A, Herring WJ. Sugammadex for Reversal of Neuromuscular Blockade in Neonates and Infants Less than 2 Years Old: Results from a Phase IV Randomized Clinical Trial. Anesthesiology. 2025 Aug 1;143(2):300-312. doi: 10.1097/ALN.0000000000005535. Epub 2025 May 5. PMID 40324166
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 145 pediatric participants between the ages of birth and <2 years undergoing a procedure requiring a neuromuscular blocking agent (NMBA) for either moderate or deep neuromuscular blockade (NMB) were enrolled in this study. Participants were enrolled in 4 age cohorts: birth to 27 days, 28 days to <3 months, 3 months to <6 months, and 6 months to <2 years.
Pre-assignment Details: 50 participants were allocated to moderate block and reversal (2 mg/kg) or deep block and reversal (4 mg/kg) with sugammadex in Part A. 95 participants were randomized in Part B to moderate block and reversal (2 mg/kg) with sugammadex, deep block and reversal (4 mg/kg) with sugammadex, or moderate block and reversal with neostigmine (50 μg/kg).
Groups:
- Part A: Sugammadex 2 mg/kg: Participants received a single intravenous (IV) bolus of sugammadex at 2 mg/kg for moderate NMB reversal.
- Part A: Sugammadex 4 mg/kg; Part B: Sugammadex 4 mg/kg: Participants received a single IV bolus of sugammadex at 4 mg/kg for deep NMB reversal.
- Part B: Sugammadex 2 mg/kg: Participants received a single IV bolus of sugammadex at 2 mg/kg for moderate NMB reversal.
- Part B: Neostigmine + (Glycopyrrolate or Atropine): Participants received a single IV bolus containing neostigmine (50 μg/kg; up to 5 mg maximum dose) in combination with either glycopyrrolate (10 μg/kg) or atropine sulfate (20 μg/kg) based on availability and/or contraindications, for moderate NMB reversal.
Period: Overall Study
Arm/Group | Part A: Sugammadex 2 mg/kg | Part A: Sugammadex 4 mg/kg | Part B: Sugammadex 2 mg/kg | Part B: Sugammadex 4 mg/kg | Part B: Neostigmine + (Glycopyrrolate or Atropine)
Started | 16 | 34 | 31 | 32 | 32
Treated | 15 | 32 | 29 | 31 | 31
Completed | 15 | 31 | 29 | 31 | 31
Not Completed | 1 | 3 | 2 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Randomized By Mistake Without Study Treatment | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal By Parent/Guardian | 0 | 2 | 1 | 1 | 0
Not completed — Previous Drug Exposure | 0 | 0 | 1 | 0 | 0
Not completed — Early Discharge | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The population used for Baseline Characteristics was the "All Participants Allocated (Part A)/Randomized (Part B) Population", with the exception of the "Protocol-defined Age Cohorts" characteristic and "Type of Neuromuscular Blocking Agent (NMBA)" Characteristic, which were reported per protocol for the "All Participants as Treated" (APaT) population.
Groups:
- Part A: Sugammadex 2 mg/kg: Participants received a single intravenous (IV) bolus of sugammadex at 2 mg/kg.
- Part A: Sugammadex 4 mg/kg; Part B: Sugammadex 4 mg/kg: Participants received a single IV bolus of sugammadex at 4 mg/kg.
- Part B: Sugammadex 2 mg/kg: Participants received a single IV bolus of sugammadex at 2 mg/kg.
- Part B: Neostigmine + (Glycopyrrolate or Atropine): Participants received a single IV bolus containing neostigmine (50 μg/kg; up to 5 mg maximum dose) in combination with either glycopyrrolate (10 μg/kg) or atropine sulfate (20 μg/kg) based on availability and/or contraindications.
- Total: Total of all reporting groups
Arm/Group | Part A: Sugammadex 2 mg/kg | Part A: Sugammadex 4 mg/kg | Part B: Sugammadex 2 mg/kg | Part B: Sugammadex 4 mg/kg | Part B: Neostigmine + (Glycopyrrolate or Atropine) | Total
Number analyzed (Participants) | 16 | 34 | 31 | 32 | 32 | 145
Age, Continuous [Mean (Standard Deviation); unit: days] | 195.9 (193.4) | 140.1 (121.7) | 157.9 (171.8) | 169.1 (165.5) | 174.3 (192.7) | 164.0 (166.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 5 | 11 | 12 | 48
  Male | 9 | 21 | 26 | 21 | 20 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 10 | 7 | 9 | 35
  Not Hispanic or Latino | 13 | 28 | 21 | 24 | 23 | 109
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 4 | 1 | 4 | 11
  Asian | 2 | 4 | 6 | 8 | 8 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 1 | 3
  White | 14 | 28 | 21 | 20 | 17 | 100
  More than one race | 0 | 0 | 0 | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Protocol-defined Age Cohorts (All Participants As Treated Population) [Count of Participants; unit: Participants] — Per protocol, Protocol-defined Age Cohorts were reported for the APaT Population and used as a stratification factor for statistical analyses. Population: "Protocol-defined Age Cohorts" characteristic was reported per protocol for the APaT population. A single participant assigned to the Sugammadex 2 mg/kg "3 months to <6 months age cohort" (N=2) was excluded from the APaT population due to missing IV dose information, but included in the corresponding cohort of the PK Evaluable Population (N=3).
  Participants
    number analyzed (Participants) | 15 | 32 | 29 | 31 | 31 | 138
    Birth to 27 days | 4 | 6 | 7 | 6 | 5 | 28
    28 days to < 3 months | 3 | 8 | 6 | 9 | 9 | 35
    3 months to < 6 months | 2 | 11 | 8 | 8 | 8 | 37
    6 months to < 2 years | 6 | 7 | 8 | 8 | 9 | 38
Type of Neuromuscular Blocking Agent [NMBA] (All Participants As Treated Population) [Count of Participants; unit: Participants] — Per protocol, Type of NMBA (rocuronium and vecuronium) was reported for the APaT Population and used as a stratification factor for statistical analyses. Population: "Type of Neuromuscular Blocking Agent (NMBA)" characteristic was reported per protocol for the APaT population.
  Participants
    number analyzed (Participants) | 15 | 32 | 29 | 31 | 31 | 138
    Rocuronium | 14 | 25 | 21 | 19 | 19 | 98
    Vecuronium | 1 | 7 | 8 | 12 | 12 | 40
EudraCT Age Categories [Count of Participants; unit: Participants] — EMA pre-defined age categories that are part of the Clinical Trial Application (CTA).
  Participants
    Newborns (0-27 days) | 4 | 6 | 7 | 6 | 6 | 29
    Infants and toddlers (28 days-23 months) | 12 | 28 | 24 | 26 | 26 | 116

OUTCOME MEASURES:

1. Primary Outcome: Part A: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC0-inf) for Sugammadex
Description: Pharmacokinetic (PK) blood samples were collected in Part A from pediatric participants at multiple collection times post administration of sugammadex using a sparse sampling approach and used to determine AUC0-inf for sugammadex. As pre-specified by the Statistical Analysis Plan (SAP) for the PK analysis, all PK parameters were analyzed and reported by Part A age cohort (birth to <27 days, 28 days to <3 months, 3 to <6 months, and 6 months to < 2 years) for each dose (2 mg and 4 mg).
Time Frame: Day 1: 2, 15, 30, 60, 240 to 360, and 600 to 720 minutes post-dose
Population: All pediatric participants in Part A who received at least 1 dose of sugammadex and had at least 5 samples at the time points of interest were analyzed per protocol by age cohort. One participant in the Sugammadex 2 mg/kg "3 months to <6 months age cohort" was evaluated for PK but excluded from the APaT population due to missing IV dose information. Per protocol, Part B participants were not analyzed for PK.
Measure: Geometric Mean (95% Confidence Interval); unit: Hour (hr)*ug/mL
Groups:
- Part A: Sugammadex 2 mg/kg [Birth to 27 Days]: Participants aged birth to 27 days received a single IV bolus of sugammadex at 2 mg/kg for moderate NMB reversal.
- Part A: Sugammadex 2 mg/kg [28 Days to <3 Months]: Participants aged 28 days to <3 months received a single IV bolus of sugammadex at 2 mg/kg for moderate NMB reversal.
- Part A: Sugammadex 2 mg/kg [3 to < 6 Months]: Participants aged 3 to < 6 months received a single IV bolus of sugammadex at 2 mg/kg for moderate NMB reversal.
- Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years]: Participants aged 6 months to < 2 years received a single IV bolus of sugammadex at 2 mg/kg for moderate NMB reversal.
- Part A: Sugammadex 4 mg/kg [Birth to 27 Days]: Participants aged birth to 27 days received a single IV bolus of sugammadex at 4 mg/kg for deep NMB reversal.
- Part A: Sugammadex 4 mg/kg [28 Days to <3 Months]: Participants aged 28 days to <3 months received a single IV bolus of sugammadex at 4 mg/kg for deep NMB reversal.
- Part A: Sugammadex 4 mg/kg [3 to < 6 Months]: Participants aged 3 to < 6 months received a single IV bolus of sugammadex at 4 mg/kg for deep NMB reversal.
- Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]: Participants aged 6 months to < 2 years received a single IV bolus of sugammadex at 4 mg/kg for deep NMB reversal.
Arm/Group | Part A: Sugammadex 2 mg/kg [Birth to 27 Days] | Part A: Sugammadex 2 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 2 mg/kg [3 to < 6 Months] | Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years] | Part A: Sugammadex 4 mg/kg [Birth to 27 Days] | Part A: Sugammadex 4 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 4 mg/kg [3 to < 6 Months] | Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 6 | 6 | 8 | 5
Hour (hr)*ug/mL | 13.40 [NA to NA] — NA = 95% confidence interval (CI) was not estimated for n<3 due to insufficient data to support its protocol pre-specified calculation. | 16.22 [12.14 to 21.67] | 11.50 [8.61 to 15.37] | 14.07 [11.24 to 17.61] | 39.09 [31.85 to 47.98] | 31.90 [25.99 to 39.16] | 24.75 [20.73 to 29.56] | 27.75 [22.17 to 34.74]
Statistical Analysis 1: Comparison: Part A: Sugammadex 2 mg/kg [Birth to 27 Days] vs Part A: Sugammadex 2 mg/kg [28 Days to <3 Months]; 2 mg/kg AUC0-inf Geometric Mean Ratio (GMR) = Birth to 27 days AUC0-inf Geometric Mean (GM) / 28 days to < 3 months AUC0-inf GM; Test type: Other; Geometric Mean Ratio (GMR) = 0.83, 90% CI 2-sided [0.56 to 1.21]
Statistical Analysis 2: Comparison: Part A: Sugammadex 2 mg/kg [28 Days to <3 Months] vs Part A: Sugammadex 2 mg/kg [3 to < 6 Months]; 2 mg/kg AUC0-inf GMR = 28 days to < 3 months AUC0-inf GM / 3 to < 6 months AUC0-inf GM; Test type: Other; Geometric Mean Ratio (GMR) = 1.41, 90% CI 2-sided [1.00 to 1.98]
Statistical Analysis 3: Comparison: Part A: Sugammadex 2 mg/kg [3 to < 6 Months] vs Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years]; 2 mg/kg AUC0-inf GMR = 3 to < 6 months AUC0-inf GM / 6 months to < 2 years AUC0-inf GM; Test type: Other; Geometric Mean Ratio (GMR) = 0.82, 90% CI 2-sided [0.60 to 1.11]
Statistical Analysis 4: Comparison: Part A: Sugammadex 4 mg/kg [Birth to 27 Days] vs Part A: Sugammadex 4 mg/kg [28 Days to <3 Months]; 4 mg/kg AUC0-inf GMR = Birth to 27 days AUC0-inf GM / 28 days to < 3 months AUC0-inf GM; Test type: Other; Geometric Mean Ratio (GMR) = 1.23, 90% CI 2-sided [0.96 to 1.56]
Statistical Analysis 5: Comparison: Part A: Sugammadex 4 mg/kg [28 Days to <3 Months] vs Part A: Sugammadex 4 mg/kg [3 to < 6 Months]; 4 mg/kg AUC0-inf GMR = 28 days to < 3 months AUC0-inf GM / 3 to < 6 months AUC0-inf GM; Test type: Other; Geometric Mean Ratio (GMR) = 1.29, 90% CI 2-sided [1.03 to 1.62]
Statistical Analysis 6: Comparison: Part A: Sugammadex 4 mg/kg [3 to < 6 Months] vs Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]; 4 mg/kg AUC0-inf GMR = 3 to < 6 months AUC0-inf GM / 6 months to < 2 years AUC0-inf GM; Test type: Other; Geometric Mean Ratio (GMR) = 0.89, 90% CI 2-sided [0.70 to 1.13]

2. Primary Outcome: Part A: Area Under the Plasma Concentration Time Curve up to the Interpolated Concentration at 1 Hour Post Dose (AUC0-1hr) for Sugammadex
Description: PK blood samples were collected in Part A from pediatric participants at multiple collection times post administration of sugammadex using a sparse sampling approach and used to determine AUC0-1hr for sugammadex. As pre-specified by the SAP for the PK analysis, all PK parameters were analyzed and reported by Part A age cohort (birth to <27 days, 28 days to <3 months, 3 to <6 months, and 6 months to < 2 years) for each dose (2 mg and 4 mg).
Time Frame: Day 1: 2, 15, 30, and 60 minutes (1 hour) post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ug/mL
Arm/Group | Part A: Sugammadex 2 mg/kg [Birth to 27 Days] | Part A: Sugammadex 2 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 2 mg/kg [3 to < 6 Months] | Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years] | Part A: Sugammadex 4 mg/kg [Birth to 27 Days] | Part A: Sugammadex 4 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 4 mg/kg [3 to < 6 Months] | Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 7 | 9 | 7
hr*ug/mL | 6.95 [5.38 to 8.99] | 7.63 [5.90 to 9.87] | 6.10 [4.72 to 7.88] | 7.31 [6.09 to 8.76] | 12.38 [10.33 to 14.85] | 14.39 [12.16 to 17.02] | 13.46 [11.61 to 15.61] | 13.92 [11.76 to 16.46]
Statistical Analysis 1: Comparison: Part A: Sugammadex 2 mg/kg [Birth to 27 Days] vs Part A: Sugammadex 2 mg/kg [28 Days to <3 Months]; 2 mg/kg AUC0-1hr GMR = Birth to 27 days AUC0-1hr GM / 28 days to < 3 months AUC0-1hr GM; Test type: Other; Geometric Mean Ratio (GMR) = 0.91, 90% CI 2-sided [0.67 to 1.23]
Statistical Analysis 2: Comparison: Part A: Sugammadex 2 mg/kg [28 Days to <3 Months] vs Part A: Sugammadex 2 mg/kg [3 to < 6 Months]; 2 mg/kg AUC0-1hr GMR = 28 days to < 3 months AUC0-1hr GM / 3 to < 6 months AUC0-1hr GM; Test type: Other; Geometric Mean Ratio (GMR) = 1.25, 90% CI 2-sided [0.92 to 1.69]
Statistical Analysis 3: Comparison: Part A: Sugammadex 2 mg/kg [3 to < 6 Months] vs Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years]; 2 mg/kg AUC0-1hr GMR = 3 to < 6 months AUC0-1hr GM / 6 months to < 2 years AUC0-1hr GM; Test type: Other; Geometric Mean Ratio (GMR) = 0.83, 90% CI 2-sided [0.64 to 1.08]
Statistical Analysis 4: Comparison: Part A: Sugammadex 4 mg/kg [Birth to 27 Days] vs Part A: Sugammadex 4 mg/kg [28 Days to <3 Months]; 4 mg/kg AUC0-1hr GMR = Birth to 27 days AUC0-1hr GM / 28 days to < 3 months AUC0-1hr GM; Test type: Other; Geometric Mean Ratio (GMR) = 0.86, 90% CI 2-sided [0.70 to 1.06]
Statistical Analysis 5: Comparison: Part A: Sugammadex 4 mg/kg [28 Days to <3 Months] vs Part A: Sugammadex 4 mg/kg [3 to < 6 Months]; 4 mg/kg AUC0-1hr GMR = 28 days to < 3 months AUC0-1hr GM / 3 to < 6 months AUC0-1hr GM; Test type: Other; Geometric Mean Ratio (GMR) = 1.07, 90% CI 2-sided [0.89 to 1.29]
Statistical Analysis 6: Comparison: Part A: Sugammadex 4 mg/kg [3 to < 6 Months] vs Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]; 4 mg/kg AUC0-1hr GMR = 3 to < 6 months AUC0-1hr GM / 6 months to < 2 years AUC0-1hr GM; Test type: Other; Geometric Mean Ratio (GMR) = 0.97, 90% CI 2-sided [0.80 to 1.17]

3. Primary Outcome: Part A: Area Under the Plasma Concentration Time Curve up to the Interpolated Concentration at 4 Hours Post Dose (AUC0-4hr) for Sugammadex
Description: PK blood samples were collected in Part A from pediatric participants at multiple collection times post administration of sugammadex using a sparse sampling approach and used to determine AUC0-4hr for sugammadex. As pre-specified by the SAP for the PK analysis, all PK parameters were analyzed and reported by Part A age cohort (birth to <27 days, 28 days to <3 months, 3 to <6 months, and 6 months to < 2 years) for each dose (2 mg and 4 mg).
Time Frame: Day 1: 2, 15, 30, 60, and 240 minutes (4 hours) post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ug/mL
Arm/Group | Part A: Sugammadex 2 mg/kg [Birth to 27 Days] | Part A: Sugammadex 2 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 2 mg/kg [3 to < 6 Months] | Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years] | Part A: Sugammadex 4 mg/kg [Birth to 27 Days] | Part A: Sugammadex 4 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 4 mg/kg [3 to < 6 Months] | Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 6 | 6 | 8 | 6
hr*ug/mL | 10.68 [NA to NA] — NA = 95% confidence interval (CI) was not estimated for n<3 due to insufficient data to support its protocol pre-specified calculation. | 13.99 [10.67 to 18.33] | 10.13 [7.73 to 13.27] | 12.57 [10.19 to 15.50] | 27.79 [22.95 to 33.64] | 27.16 [22.43 to 32.89] | 21.51 [18.23 to 25.39] | 22.43 [18.52 to 27.15]

4. Primary Outcome: Part A: Maximum Plasma Concentration (Cmax) of Sugammadex
Description: PK blood samples were collected in Part A from pediatric participants at multiple collection times post administration of sugammadex using a sparse sampling approach and used to determine Cmax for sugammadex. As pre-specified by the SAP for the PK analysis, all PK parameters were analyzed and reported by Part A age cohort (birth to <27 days, 28 days to <3 months, 3 to <6 months, and 6 months to < 2 years) for each dose (2 mg and 4 mg).
Time Frame: Day 1: 2, 15, 30, 60, 240 to 360, and 600 to 720 minutes post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Part A: Sugammadex 2 mg/kg [Birth to 27 Days] | Part A: Sugammadex 2 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 2 mg/kg [3 to < 6 Months] | Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years] | Part A: Sugammadex 4 mg/kg [Birth to 27 Days] | Part A: Sugammadex 4 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 4 mg/kg [3 to < 6 Months] | Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 6 | 8 | 9 | 7
ug/mL | 19.59 [14.15 to 27.13] | 21.18 [14.55 to 30.84] | 19.39 [13.32 to 28.23] | 20.99 [16.09 to 27.38] | 28.56 [21.89 to 37.25] | 30.38 [24.13 to 38.24] | 44.51 [35.83 to 55.29] | 40.86 [31.95 to 52.25]
Statistical Analysis 1: Comparison: Part A: Sugammadex 2 mg/kg [Birth to 27 Days] vs Part A: Sugammadex 2 mg/kg [28 Days to <3 Months]; 2 mg/kg Cmax GMR = Birth to 27 days Cmax GM / 28 days to < 3 months Cmax GM; Test type: Other; Geometric Mean Ratio (GMR) = 0.92, 90% CI 2-sided [0.61 to 1.40]
Statistical Analysis 2: Comparison: Part A: Sugammadex 2 mg/kg [28 Days to <3 Months] vs Part A: Sugammadex 2 mg/kg [3 to < 6 Months]; 2 mg/kg Cmax GMR = 28 days to < 3 months Cmax GM / 3 to < 6 months Cmax GM; Test type: Other; Geometric Mean Ratio (GMR) = 1.09, 90% CI 2-sided [0.70 to 1.70]
Statistical Analysis 3: Comparison: Part A: Sugammadex 2 mg/kg [3 to < 6 Months] vs Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years]; 2 mg/kg Cmax GMR = 3 to < 6 months Cmax GM / 6 months to < 2 years Cmax GM; Test type: Other; Geometric Mean Ratio (GMR) = 0.92, 90% CI 2-sided [0.63 to 1.36]
Statistical Analysis 4: Comparison: Part A: Sugammadex 4 mg/kg [Birth to 27 Days] vs Part A: Sugammadex 4 mg/kg [28 Days to <3 Months]; 4 mg/kg Cmax GMR = Birth to 27 days Cmax GM / 28 days to < 3 months Cmax GM; Test type: Other; Geometric Mean Ratio (GMR) = 0.94, 90% CI 2-sided [0.70 to 1.26]
Statistical Analysis 5: Comparison: Part A: Sugammadex 4 mg/kg [28 Days to <3 Months] vs Part A: Sugammadex 4 mg/kg [3 to < 6 Months]; 4 mg/kg Cmax GMR = 28 days to < 3 months Cmax GM / 3 to < 6 months Cmax GM; Test type: Other; Geometric Mean Ratio (GMR) = 0.68, 90% CI 2-sided [0.52 to 0.89]
Statistical Analysis 6: Comparison: Part A: Sugammadex 4 mg/kg [3 to < 6 Months] vs Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]; 4 mg/kg AUC0-1hr GMR = 3 to < 6 months Cmax GM / 6 months to < 2 years Cmax GM; Test type: Other; Geometric Mean Ratio (GMR) = 1.09, 90% CI 2-sided [0.83 to 1.43]

5. Primary Outcome: Part A: Plasma Clearance (CL) of Sugammadex
Description: PK blood samples were collected in Part A from pediatric participants at multiple collection times post administration of sugammadex using a sparse sampling approach and used to determine CL for sugammadex. As pre-specified by the SAP for the PK analysis, all PK parameters were analyzed and reported by Part A age cohort (birth to <27 days, 28 days to <3 months, 3 to <6 months, and 6 months to < 2 years) for each dose (2 mg and 4 mg).
Time Frame: Day 1: 2, 15, 30, 60, 240 to 360, and 600 to 720 minutes post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Liters/hour
Arm/Group | Part A: Sugammadex 2 mg/kg [Birth to 27 Days] | Part A: Sugammadex 2 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 2 mg/kg [3 to < 6 Months] | Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years] | Part A: Sugammadex 4 mg/kg [Birth to 27 Days] | Part A: Sugammadex 4 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 4 mg/kg [3 to < 6 Months] | Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 6 | 6 | 8 | 5
Liters/hour | 0.43 [NA to NA] — NA = 95% confidence interval (CI) was not estimated for n<3 due to insufficient data to support its protocol pre-specified calculation. | 0.66 [0.47 to 0.92] | 1.28 [0.91 to 1.80] | 1.34 [1.03 to 1.74] | 0.35 [0.28 to 0.45] | 0.61 [0.48 to 0.78] | 0.97 [0.79 to 1.19] | 1.27 [0.98 to 1.65]

6. Primary Outcome: Part A: Apparent Volume of Distribution (Vd) for Sugammadex
Description: PK blood samples were collected in Part A from pediatric participants at multiple collection times post administration of sugammadex using a sparse sampling approach and used to determine Vd for sugammadex. As pre-specified by the SAP for the PK analysis, all PK parameters were analyzed and reported by Part A age cohort (birth to <27 days, 28 days to <3 months, 3 to <6 months, and 6 months to < 2 years) for each dose (2 mg and 4 mg).
Time Frame: Day 1: 2, 15, 30, 60, 240 to 360, and 600 to 720 minutes post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Liters (L)
Arm/Group | Part A: Sugammadex 2 mg/kg [Birth to 27 Days] | Part A: Sugammadex 2 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 2 mg/kg [3 to < 6 Months] | Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years] | Part A: Sugammadex 4 mg/kg [Birth to 27 Days] | Part A: Sugammadex 4 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 4 mg/kg [3 to < 6 Months] | Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 6 | 6 | 8 | 5
Liters (L) | 1.14 [NA to NA] — NA = 95% confidence interval (CI) was not estimated for n<3 due to insufficient data to support its protocol pre-specified calculation. | 1.45 [1.06 to 1.98] | 2.68 [1.96 to 3.67] | 2.70 [2.11 to 3.44] | 1.22 [0.98 to 1.52] | 1.35 [1.08 to 1.68] | 2.16 [1.78 to 2.62] | 2.77 [2.17 to 3.53]

7. Primary Outcome: Apparent Volume of Distribution at Steady State (Vss) for Sugammadex
Description: PK blood samples were collected in Part A from pediatric participants at multiple collection times post administration of sugammadex using a sparse sampling approach and used to determine Vss for sugammadex. As pre-specified by the SAP for the PK analysis, all PK parameters were analyzed and reported by Part A age cohort (birth to <27 days, 28 days to <3 months, 3 to <6 months, and 6 months to < 2 years) for each dose (2 mg and 4 mg).
Time Frame: Day 1: 2, 15, 30, 60, 240 to 360, and 600 to 720 minutes post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Liters (L)
Arm/Group | Part A: Sugammadex 2 mg/kg [Birth to 27 Days] | Part A: Sugammadex 2 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 2 mg/kg [3 to < 6 Months] | Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years] | Part A: Sugammadex 4 mg/kg [Birth to 27 Days] | Part A: Sugammadex 4 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 4 mg/kg [3 to < 6 Months] | Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 6 | 6 | 8 | 5
Liters (L) | 1.04 [NA to NA] — NA = 95% confidence interval (CI) was not estimated for n<3 due to insufficient data to support its protocol pre-specified calculation. | 1.23 [0.94 to 1.60] | 2.07 [1.59 to 2.70] | 2.14 [1.74 to 2.63] | 1.11 [0.92 to 1.34] | 1.18 [0.98 to 1.43] | 1.69 [1.43 to 1.98] | 2.18 [1.77 to 2.68]

8. Primary Outcome: Part A: Half-Life (t1/2) of Sugammadex in Plasma
Description: PK blood samples were collected in Part A from pediatric participants at multiple collection times post administration of sugammadex using a sparse sampling approach and used to determine t½ for sugammadex. As pre-specified by the SAP for the PK analysis, all PK parameters were analyzed and reported by Part A age cohort (birth to <27 days, 28 days to <3 months, 3 to <6 months, and 6 months to < 2 years) for each dose (2 mg and 4 mg).
Time Frame: Day 1: 2, 15, 30, 60, 240 to 360, and 600 to 720 minutes post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | Part A: Sugammadex 2 mg/kg [Birth to 27 Days] | Part A: Sugammadex 2 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 2 mg/kg [3 to < 6 Months] | Part A: Sugammadex 2 mg/kg [6 Months to < 2 Years] | Part A: Sugammadex 4 mg/kg [Birth to 27 Days] | Part A: Sugammadex 4 mg/kg [28 Days to <3 Months] | Part A: Sugammadex 4 mg/kg [3 to < 6 Months] | Part A: Sugammadex 4 mg/kg [6 Months to < 2 Years]
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 6 | 6 | 9 | 5
Hours (h) | 1.84 (NA) — NA = 95% confidence interval (CI) was not estimated for n<3 due to insufficient data to support its protocol pre-specified calculation. | 1.52 (20.21) | 1.45 (28.57) | 1.40 (24.25) | 2.39 (27.34) | 1.53 (16.42) | 1.51 (28.79) | 1.51 (19.46)

9. Primary Outcome: Part B: Time to Neuromuscular Recovery (TTNMR) In Reversal of Moderate Block
Description: Time to neuromuscular recovery was defined as the interval from administration of reversal agent to time to neuromuscular recovery. TTNMR could be assessed by 1 of 4 methods selected by the investigator, based on their judgment of what was technically feasible and clinically appropriate for the participant's procedure. These methods were inclusive of both clinical signs (head lift or hip flexion) and neuromuscular transmission monitoring using either a standard peripheral nerve stimulator or the technically challenging quantitative neuromuscular monitoring to train-of-four (TOF) ratio ≥0.9. As pre-specified by the protocol and SAP, TTNMR was analyzed only in Part B participants under the setting of moderate block for comparison of sugammadex 2 mg to neostigmine.
Time Frame: Within Day 1
Population: All randomized participants in Part B who received ≥1 dose of study treatment for moderate NMB reversal (i.e. Sugammadex 2 mg/kg or Neostigmine + [Glycopyrrolate or Atropine]) and with available TTNMR data were analyzed. Per the protocol objective, no formal test for efficacy with comparison to neostigmine was done for Part A and Part B deep block, thus Part A and Part B 4 mg/kg participants were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Part A: Sugammadex 2 mg/kg | Part A: Sugammadex 4 mg/kg | Part B: Sugammadex 2 mg/kg | Part B: Sugammadex 4 mg/kg | Part B: Neostigmine + (Glycopyrrolate or Atropine)
Number analyzed (Participants) | 0 | 0 | 29 | 0 | 31
Minutes |  |  | 1.4 (1.1) [1.1 to 2.0] |  | 4.4 (2.7) [2.7 to 7.9]
Statistical Analysis 1: Comparison: Part B: Sugammadex 2 mg/kg vs Part B: Neostigmine + (Glycopyrrolate or Atropine); The Hazard Ratio (HR) for the pairwise comparison of Sugammadex 2 mg/kg vs. Neostigmine + (Glycopyrrolate or Atropine) was based on a Cox regression model with Efron's method of tie handling with covariates of treatment, age (continuous) and stratified by neuromuscular blocking agent; Test type: Superiority; p = 0.0002, Log Rank — Two-sided p-value based on log-rank test stratified by neuromuscular blocking agent and age groups; Hazard Ratio (HR) = 2.40, 95% CI 2-sided [1.37 to 4.18]

10. Primary Outcome: Parts A and B: Percentage of Participants With Adverse Events (AEs) Up To 7 Days Post Administration of Study Medication
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. As pre-specified by the protocol and SAP, the primary analysis of safety combined data across Part A and Part B (and across age cohorts) and included all AEs that occurred up to 7 days post administration of study medication. The percentage of participants with an AE was reported by treatment and dose received.
Time Frame: Up to Day 7
Population: All enrolled/randomized participants from both Part A and Part B (combined per protocol) who received at least 1 dose of study treatment were analyzed.
Measure: Number; unit: Percentage of Participants
Groups:
- Parts A + B: Sugammadex 2 mg/kg: Participants in Parts A and B received a single IV bolus of sugammadex at 2 mg/kg for moderate NMB reversal.
- Parts A + B: Sugammadex 4 mg/kg: Participants in Parts A and B received a single IV bolus of sugammadex at 4 mg/kg for deep NMB reversal.
Arm/Group | Parts A + B: Sugammadex 2 mg/kg | Parts A + B: Sugammadex 4 mg/kg | Part B: Neostigmine + (Glycopyrrolate or Atropine)
Number analyzed (Participants) | 44 | 63 | 31
Percentage of Participants | 68.2 | 68.3 | 61.3
Statistical Analysis 1: Comparison: Parts A + B: Sugammadex 2 mg/kg vs Part B: Neostigmine + (Glycopyrrolate or Atropine); The difference in percentage of participants with an AE in sugammadex 2 mg/kg group versus the Neostigmine + (Glycopyrrolate or Atropine) group was based on the Miettinen and Nurminen method stratified by neuromuscular blocking agent and age group; Test type: Other; Difference in Percentage = 7.6, 95% CI 2-sided [-14.2 to 29.5]
Statistical Analysis 2: Comparison: Parts A + B: Sugammadex 4 mg/kg vs Part B: Neostigmine + (Glycopyrrolate or Atropine); The difference in percentage of participants with an AE in sugammadex 4 mg/kg group versus the Neostigmine + (Glycopyrrolate or Atropine) group was based on the Miettinen and Nurminen method stratified by neuromuscular blocking agent and age group; Test type: Other; Difference in Percentage = 5.9, 95% CI 2-sided [-13.5 to 26.7]

11. Secondary Outcome: Part B: Time to Extubation In Reversal of Moderate Block
Description: Time to extubation was defined as the interval from administration of reversal agent to removal of the endotracheal tube. Monitoring of time to extubation during Part B (moderate block) was achieved using the Extubation Readiness Assessment, which evaluated and documented clinically relevant elements including neuromuscular recovery, mental status, return of spontaneous ventilation, adequate oxygenation, hemodynamically stabile, and core body temperature with "Yes"/"No" answers (no overall score or direction attributed). The Operating Room anesthesiologist or other trained personnel were responsible for assessing extubation readiness beginning about 1 minute after study treatment administration and reassessing every 60 seconds until time of extubation readiness was achieved. As pre-specified by the protocol, Time to Extubation was analyzed only in Part B under setting of moderate block, and Part A participants were not included in this analysis.
Time Frame: Within Day 1
Population: All randomized participants in Part B who received ≥1 dose of study treatment for moderate NMB reversal (i.e. Sugammadex 2 mg/kg or Neostigmine + [Glycopyrrolate or Atropine]) were analyzed. Per the protocol objective, no formal test for efficacy with comparison to neostigmine was done for Part A and Part B deep block, thus Part A and Part B 4 mg/kg participants were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Part A: Sugammadex 2 mg/kg | Part A: Sugammadex 4 mg/kg | Part B: Sugammadex 2 mg/kg | Part B: Sugammadex 4 mg/kg | Part B: Neostigmine + (Glycopyrrolate or Atropine)
Number analyzed (Participants) | 0 | 0 | 29 | 0 | 31
Minutes |  |  | 7.9 (5.7) [5.7 to 11.6] |  | 10.5 (7.9) [7.9 to 13.5]

ADVERSE EVENTS:
Time Frame: Up to Day 14
Description: All-Cause Mortality includes all allocated (Part A)/randomized (Part B) participants. Serious adverse events (SAEs) and Nonserious AEs include all allocated/randomized participants who received ≥1 dose of study drug.
Arm/Group | Part A: Sugammadex 2 mg/kg | Part A: Sugammadex 4 mg/kg | Part B: Sugammadex 2 mg/kg | Part B: Sugammadex 4 mg/kg | Part B: Neostigmine + (Glycopyrrolate or Atropine)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/34 | 0/31 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/32 | 3/29 | 1/31 | 0/31
Other Adverse Events (participants affected / at risk) | 11/15 | 22/32 | 19/29 | 17/31 | 16/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Sugammadex 2 mg/kg (N=15) | Part A: Sugammadex 4 mg/kg (N=32) | Part B: Sugammadex 2 mg/kg (N=29) | Part B: Sugammadex 4 mg/kg (N=31) | Part B: Neostigmine + (Glycopyrrolate or Atropine) (N=31)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device mechanical issue (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Sugammadex 2 mg/kg (N=15) | Part A: Sugammadex 4 mg/kg (N=32) | Part B: Sugammadex 2 mg/kg (N=29) | Part B: Sugammadex 4 mg/kg (N=31) | Part B: Neostigmine + (Glycopyrrolate or Atropine) (N=31)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 7 (7) | 21 (22) | 11 (12) | 13 (13) | 10 (10)
Procedural vomiting (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irregular breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT03909165/Prot_SAP_000.pdf